CLINICAL TRIAL: NCT06076239
Title: Effect of ESWT Applied on the Trigger Point on Pain Function and Effusion in Individuals With Shoulder Impingement Syndrome
Brief Title: Effect of Extracorporeal Shock Wave Therapy in Impingement Syndrome
Acronym: ESWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Seçil ÖZKURT, Asst. Prof. Dr., Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5000009
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Shoulder Impingement Syndrome; Trigger Point Pain
Keywords: extracorporeal shock wave therapy; shoulder pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The participants in the Experimental Group were given Extra Corporeal Shockwave therapy to the trigger point of the patients with a trigger point in one of the supraspinatus, subscapularis and infraspinatus muscles for a total of 5 sessions in 3 weeks (2 sessions in the first week, 2 sessions in the second week, 1 session in the third week) in addition to conventional treatments , while Control group received only conventional treatments for five days per week for 3 consecutive weeks
Who Masked: Outcomes Assessor
Masking Description: Supraspinatus tendon thickness and effusion of the cases included in the study were evaluated by ultrasonography before and after the study by the same specialist physician who was blind to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT Group (Experimental): The participants in the ESWT Group (n=16) were given Extracorporeal Shock Wave Therapy to the trigger point of the patients with a trigger point in one of the supraspinatus, subscapularis and infraspinatus muscles for a total of 5 sessions in 3 weeks (2 sessions in the first week, 2 sessions in the second week, 1 session in the third week) in addition to conventional treatment.1000 pulses to the trigger point of the patients with a trigger point in one of the supraspinatus, subscapularis and infraspinatus muscles, 500 pulses to the surrounding area, 2 bars, ESWT (GYMNMA Shockmaster 500) was applied for a total of 5 sessions in 3 weeks at 10 Hz, medium energy level (<0.28 mJ/mm2).
  Interventions: Other: ESWT Group
- Control Group (Active Comparator): Control group (n=16) received only conventional treatment for five days per week for 3 consecutive weeks. Conventional treatment includes Ultrasound therapy(Gymna Pulson200) (1 mHz. treatment dose average 1.5 w/cm², intermittent with a small head (50%), 5 minutes around the glenohumeral joint of the cases in both groups participating in the study; at an intensity that the patient can tolerate, covering the painful area TENS applied (modified biphasic asymmetric pulse, and it was set to a pulse width of 100 μs and a frequency of 100 Hz, 20 min,) (Hometech ht 66b); hotpack and exercises (posterior capsule stretching, wand exercises, mobilization approximately 60 minutes of conventional treatment consisting of exercises and shoulder isometric exercises) was applied once a day, 5 times a week in both groups.
  Interventions: Other: ESWT Group; Other: Control Group

INTERVENTIONS:
Other: ESWT Group — EG were given Extracorporeal Shock Wave Therapy to the trigger point of the patients with a trigger point in one of the supraspinatus, subscapularis and infraspinatus muscles for a total of 5 sessions in 3 weeks (2 sessions in the first week, 2 sessions in the second week, 1 session in the third week) in addition to conventional treatment. 1000 pulses to the trigger point of the patients with a trigger point in one of the supraspinatus, subscapularis and infraspinatus muscles, 500 pulses to the surrounding area, 2 bars, ESWT (GYMNMA Shockmaster 500) was applied for a total of 5 sessions in 3 weeks at 10 Hz, medium energy level (<0.28 mJ/mm2).
  Other Names: EG
Other: Control Group — Both EG and CG were given conventional treatment.Conventional treatment is consist of Ultrasound therapy (Gymna Pulson200) (1 mHz. treatment dose average 1.5 w/cm², intermittent with a small head (50%), 5 minutes (45)) around the glenohumeral joint of the cases in both groups participating in the study; TENS applied at an intensity that the patient can tolerate, covering the painful area (modified biphasic asymmetric pulse, and it was set to a pulse width of 100 μs and a frequency of 100 Hz, 20 min,) (Hometech ht 66b); hotpack and exercises (posterior capsule stretching, wand exercises, mobilization approximately 60 minutes of conventional treatment consisting of exercises and shoulder isometric exercises) was applied once a day, 5 times a week in both groups.
  Other Names: CG
  Arms: Control Group

SUMMARY:
Purpose: This study aimed to investigate the effectiveness of ESWT applied to trigger points on pain, function, and effusion in individuals diagnosed with shoulder impingement syndrome.

Material and methods: This was a randomized controlled clinical trial with a total of 32 which were randomly divided into two equal groups (ESWT Group (EG), n = 16; Control Group (CG), n=16). The participants in the EG were given Extracorporeal Shock Wave Therapy to the trigger point of the patients with a trigger point in one of the supraspinatus, subscapularis and infraspinatus muscles for a total of 5 sessions in 3 weeks (2 sessions in the first week, 2 sessions in the second week, 1 session in the third week) in addition to conventional treatment while CG received only conventional treatments for five days per week for 3 consecutive weeks. The primary outcome was pain intensity Visual analog scale (VAS). Secondary measurements were Tendon thickness and effusion with Ultrasound, Range of motion (ROM), Manual muscle testing (MMT), Corbin posture analysis, Constant Murley Score (CMS), Arm Shoulder and Hand Problems Questionnaire (DASH). Supraspinatus tendon thickness and effusion of the cases included in the study were evaluated by ultrasonography before and after the treatment(3 weeks) by the same specialist physician who was blind to the groups. Normal joint range of motion by universal goniometer, muscle strength by manual muscle test, posture evaluation by Corbin posture analysis, pain evaluation by Visual Analogue Scale (VAS), functional evaluation by Constant Murley Score (CMS), Arm Shoulder and Hand Problems Questionnaire (DASH) by physiotherapist It was evaluated before and after the treatment (3 weeks).

DETAILED DESCRIPTION:
This study aimed to investigate the effectiveness of ESWT applied to trigger points on pain, function, and effusion in individuals diagnosed with shoulder impingement syndrome.

This was a randomized controlled clinical trial with a total of 32 which were randomly divided into two equal groups (ESWT Group (EG), n = 16; Control Group (CG), n=16). The participants in the EG were given Extracorporeal Shock Wave Therapy to the trigger point of the patients with a trigger point in one of the supraspinatus, subscapularis and infraspinatus muscles for a total of 5 sessions in 3 weeks (2 sessions in the first week, 2 sessions in the second week, 1 session in the third week) in addition to conventional treatments , while CG received only conventional treatment for five days per week for 3 consecutive weeks. Conventional treatment consist of Ultrasound treatment (Gymna Pulson200) (1 mHz. treatment dose average 1.5 w/cm², intermittent with a small head (50%), 5 minutes ) around the glenohumeral joint of the cases in both groups participating in the study; at an intensity that the patient can tolerate, covering the painful area TENS (modified biphasic asymmetric pulse, and it was set to a pulse width of 100 μs and a frequency of 100 Hz, 20 min,) (Hometech ht 66b) applied; hotpack and exercises (posterior capsule stretching, wand exercises, mobilization approximately 60 minutes of conventional treatment consisting of exercises and shoulder isometric exercises) was applied once a day, 5 times a week in both groups. In addition to conventional physiotherapy. additional to conventional treatment EG was applied 1000 pulses to the trigger point of the patients with a trigger point in one of the supraspinatus, subscapularis and infraspinatus muscles, 500 pulses to the surrounding area, 2 bars, ESWT (GYMNMA Shockmaster 500) was applied for a total of 5 sessions in 3 weeks (2 sessions in the first week, 2 sessions in the second week, 1 session in the third week) at 10 Hz, medium energy level (<0.28 mJ/mm2).Supraspinatus tendon thickness and effusion of the cases included in the study were evaluated by ultrasonography before and after the treatment(3 weeks) by the same specialist physician who was blind to the groups. Normal joint range of motion by universal goniometer, muscle strength by manual muscle test, posture evaluation by Corbin posture analysis, pain evaluation by Visual Analogue Scale (VAS), functional evaluation by Constant Murley Score (CMS), Arm Shoulder and Hand Problems Questionnaire (DASH) by physiotherapist It was evaluated before and after the treatment (3 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Having an active trigger point in the infraspinatus, supraspinatus, subscapularis muscles.
* Positive impingement tests such as Hawkings, Neer and Jobe test, 60°-120° painful arc of motion are positive.
* who were diagnosed with impingement syndrome by ultrasonography (USG) and clinical examination.

Exclusion Criteria:

* patients with severe dementia or psychiatric disease,
* diabetic patients with sensory problems,
* and a history of malignancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 3 week
  The Visual Analog Scale that is highly feasible for clinical research and practice to assess pain intensity was scored by means of a 10-cm long horizontal line ranging from (0 cm = no pain) at one end to (10 cm = maximum imaginable pain) at the other on which participants marked a point according to their subjective perception of pain

SECONDARY OUTCOMES:
Thickness of supraspinatus tendon | 3 week
  Ultrasound is a reliable method of assessing the thickness of the tendon and having the advantages of being readily available, highly sensitive, relatively inexpensive, and non-invasive. The settings of the US system were standardized for all participants and remained the same for all measurements.
Effusion in shoulder | 3 week
  Ultrasound is a reliable method of assessing the thickness of the tendon and having the advantages of being readily available, highly sensitive, relatively inexpensive, and non-invasive. The settings of the US system were standardized for all participants and remained the same for all measurements.
Shoulder ROM (flexion,extension,abduction,adduction,internal rotation,external rotation) | 3 week
  The standard (universal) goniometer that is low cost, affordable, easy to be employed measurement tool to measure for range of motion in clinical evaluations of patients (33, 34). Universal 31-centimeter plastic 180° goniometer was used
Shoulder muscle strength | 3 week
  The manual muscle test (MMT) is a flexible diagnostic tool, which is used to assess muscle strength, a "muscle power function" according to the International Classification of Functioning, Disability, and Health is defined herein as the maximum voluntary resultant output that muscles can bring to bear on the environment under a specific set of test conditions (35). 6-degree scale ranging from palsy ("Gone-no contraction felt") up to full power ("normal-muscle can hold the test position against strong pressure''
Corbin posture analyze | 3 week
  Corbin Posture Analysis is a method in which postural changes are analyzed by observing the patient's current position. Analyzes are performed from lateral and posterior perspectives, and posture is scored according to the severity of the abnormality (0 = none, 1 = mild, 2 = moderate, 3 = severe). Postural scores obtained by posterior and lateral observation are summed and graded as poor ≥12, fair 8-11, good 5-7, very good 3-4 and excellent 0-2.
Constant Murley Score | 3 week
  The CMS is a standardized, a relatively unique, simple clinical method of assessing shoulder function and has a maximum score of 100 points, with both subjective (35 points) and objective (65 points) components for various shoulder pathologies (38). The subjective parameters assess the degree of pain perception (15 points) and the ability to perform the normal tasks of daily living in both activity- and position-related terms (20 points). The objective parameters include testing of active range of motion (40 points) and muscle strength (25 points). The calculation of the score is simple and easy. A higher score corresponds to better shoulder function.
DASH | 3 week
  The Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire is the most commonly applied patient-reported outcome measure used to measure physical, psychological and social role function in clinical research and practice for patients with injuries and diseases of the upper extremities. The main component of the DASH is a 30-item scale concerning the patient's health status during the preceding week: 21 items regarding the degree of difficulty in performing certain physical activities; five items pertaining to the severity of pain, activity-related pain, tingling, weakness, and stiffness; and four items concerning the effect that the upper limb problem has had on social activities, work, sleep, and self-image. Each item is scored on a five-point ordinal scale. the DASH score results are inverted with the higher scores (maximum = 100) representing a greater disability and the lower scores occurring in a good functioning arm

CONTACTS AND LOCATIONS:
Overall Officials: Seçil Özkurt, Phd, Study Director — İstanbul Arel University
Locations (1):
- Private Olympos Hospital, Antalya, Turkey (Türkiye)